CLINICAL TRIAL: NCT03951649
Title: Acute Headache Treatment in Pregnancy: Improvement in Pain Scores With Occipital Nerve Block vs PO Acetaminophen With Caffeine A Randomized Controlled Trial
Brief Title: Acute Headache Treatment in Pregnancy: Occipital Nerve Block vs PO Acetaminophen With Caffeine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachel Sinkey, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA123456789
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Headache; Pregnancy Related; Occipital Nerve Block
Keywords: headache; Pregnancy; Acute treatment; Emergency department; Occipital nerve block
MeSH Terms: conditions — Headache; Emergencies | interventions — Acetaminophen; Caffeine

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trail
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Occipital Nerve block (Experimental): 1. Trained OB/GYN providers will perform a physical exam to access location of occipital nerve injection based on palpation of bony landmarks.
  2. Site of injection will be cleaned with an alcohol swab.
  3. 5cc of 0.5% bupivacaine will be injected into both right and left occipital nerves using a 2.5 inch 25 gauge needle. The needle will be changed between injecting sites.
  4. After injection is completed sterile gauze will be held on injection sites for 2-3 min or until bleeding is resolved.
  Interventions: Drug: Occipital Nerve Block
- Oral Acetaminophen/Caffeine Group (Active Comparator): Acetaminophen 650mg PO and Caffeine 100mg PO (both Level A treatments for acute headache)
  Interventions: Drug: Occipital Nerve Block

INTERVENTIONS:
Drug: Occipital Nerve Block — This is an open label randomized controlled trial evaluating response to bupivacaine occipital nerve block compared to Tylenol/Caffeine cocktail in treatment of pregnant patients seeking care of headache.
  Other Names: Acetaminophen/Caffeine

SUMMARY:
This is an open label randomized controlled trial evaluating response to bupivacaine occipital nerve block compared to Tylenol/Caffeine cocktail in treatment of pregnant patients seeking care of headache.

DETAILED DESCRIPTION:
This is an open label randomized controlled trial. Women who present to the MEU with headache will be assessed by trained nurse practitioners and/or OB/GYN residents. If the woman meets criteria for the study she will be enrolled by an MEU provider doing the primary assessment.

See Figure 1 for the flow diagram depicting the patient's course through MEU. If eligible for inclusion, women will be randomly assigned to ONB or headache cocktail. Randomization will occur at time of enrollment. Prior to headache treatment 10-point visual/verbal rating scale (VRS) will be obtained. Treatment time is defined as time the patient takes the medication or the time that the needle is inserted into the greater occipital notch. At 60 min after treatment VRS will again be obtained by nursing staff or primary provider. If headache pain is resolved, defined as a VRS 0, the patient will be discharged to home (at the discretion of the managing team providing there are no other indications for further observation or admission). If pain continues to be present VRS will again be assessed at 120 min after treatment. If pain is not improved to mild range, defined as a VRS ≤ 3, or resolved, crossover treatment will be given. VRS will be obtained at 60 min after cross over treatment; if pain is resolved patient will be discharge to home. If pain continues to be present VRS will be obtained at 120 min after cross over treatment. If pain is not improved to mild pain or resolved; second line treatment of Promethazine 25mg/Benadryl 25mg will be given. VRS will again be obtained 60 min after second line treatment. If pain is not improved to mild pain (VRS ≤3) or resolved neurology consult will be considered. If at any point during treatment the patient develops new neurological symptoms study protocol will be stopped and neurology will be consulted.

Patients will be called 7 days after discharge to access short term outcomes (headache frequency since MEU visit, injection site complications, and satisfaction with treatment.) Patients will again be called at 28 days and a chart abstraction will be done to access for long term outcomes (recurrent presentation for headache to the MEU, maternal complications including preeclampsia, or fetal complications).

ELIGIBILITY:
Inclusion criteria:

1. Women presenting to Maternal Evaluation Unit at UAB hospital
2. Confirmed live intrauterine pregnancy (previous ultrasound, bedside ultrasound, fetal monitoring)
3. Complaint of headache
4. Minimal pain level of 4 on VRS

Exclusion criteria:

1. Systolic BP >= 140 or diastolic BP>=90 with 1+ protein on urine dip
2. Systolic BP >=160 or diastolic BP>=105
3. Focal neurological symptoms
4. Altered level of consciousness defined as not being oriented to person, place, situation, and/or year
5. Complaint of seizure
6. Known under lying brain abnormality
7. Fever
8. Use of >3 grams of acetaminophen in past 24hrs
9. ONB in the past 3 months
10. Reported allergy to study medications (Bupivacaine, acetaminophen, or caffeine)

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant Females
Enrollment: 62 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Women and Infants center at the University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen BK, Jensen R, Schroll M, Olesen J. Epidemiology of headache in a general population--a prevalence study. J Clin Epidemiol. 1991;44(11):1147-57. doi: 10.1016/0895-4356(91)90147-2. PMID 1941010
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Scharff L, Marcus DA, Turk DC. Headache during pregnancy and in the postpartum: a prospective study. Headache. 1997 Apr;37(4):203-10. doi: 10.1046/j.1526-4610.1997.3704203.x. PMID 9150614
- [Background] Bushman ET, Varner MW, Digre KB. Headaches Through a Woman's Life. Obstet Gynecol Surv. 2018 Mar;73(3):161-173. doi: 10.1097/OGX.0000000000000540. PMID 29595872
- [Background] Robbins MS, Farmakidis C, Dayal AK, Lipton RB. Acute headache diagnosis in pregnant women: a hospital-based study. Neurology. 2015 Sep 22;85(12):1024-30. doi: 10.1212/WNL.0000000000001954. Epub 2015 Aug 19. PMID 26291282
- [Background] Loder E, Biondi D. General principles of migraine management: the changing role of prevention. Headache. 2005 Apr;45 Suppl 1:S33-47. doi: 10.1111/j.1526-4610.2005.4501002.x. PMID 15833089
- [Background] Cuadrado ML, Aledo-Serrano A, Navarro P, Lopez-Ruiz P, Fernandez-de-Las-Penas C, Gonzalez-Suarez I, Orviz A, Fernandez-Perez C. Short-term effects of greater occipital nerve blocks in chronic migraine: A double-blind, randomised, placebo-controlled clinical trial. Cephalalgia. 2017 Aug;37(9):864-872. doi: 10.1177/0333102416655159. Epub 2016 Jun 12. PMID 27296456
- [Background] Dach F, Eckeli AL, Ferreira Kdos S, Speciali JG. Nerve block for the treatment of headaches and cranial neuralgias - a practical approach. Headache. 2015 Feb;55 Suppl 1:59-71. doi: 10.1111/head.12516. Epub 2015 Feb 3. PMID 25644836
- [Background] Gul HL, Ozon AO, Karadas O, Koc G, Inan LE. The efficacy of greater occipital nerve blockade in chronic migraine: A placebo-controlled study. Acta Neurol Scand. 2017 Aug;136(2):138-144. doi: 10.1111/ane.12716. Epub 2016 Dec 2. PMID 27910088
- [Background] Hascalovici JR, Robbins MS. Peripheral Nerve Blocks for the Treatment of Headache in Older Adults: A Retrospective Study. Headache. 2017 Jan;57(1):80-86. doi: 10.1111/head.12992. Epub 2016 Nov 30. PMID 27901275
- [Background] Tang Y, Kang J, Zhang Y, Zhang X. Influence of greater occipital nerve block on pain severity in migraine patients: A systematic review and meta-analysis. Am J Emerg Med. 2017 Nov;35(11):1750-1754. doi: 10.1016/j.ajem.2017.08.027. Epub 2017 Aug 14. PMID 28844531
- [Background] Tobin J, Flitman S. Occipital nerve blocks: when and what to inject? Headache. 2009 Nov-Dec;49(10):1521-33. doi: 10.1111/j.1526-4610.2009.01493.x. Epub 2009 Aug 6. PMID 19674126
- [Background] Blumenfeld A, Ashkenazi A, Napchan U, Bender SD, Klein BC, Berliner R, Ailani J, Schim J, Friedman DI, Charleston L 4th, Young WB, Robertson CE, Dodick DW, Silberstein SD, Robbins MS. Expert consensus recommendations for the performance of peripheral nerve blocks for headaches--a narrative review. Headache. 2013 Mar;53(3):437-46. doi: 10.1111/head.12053. Epub 2013 Feb 13. PMID 23406160
- [Background] Voigt CL, Murphy MO. Occipital nerve blocks in the treatment of headaches: safety and efficacy. J Emerg Med. 2015 Jan;48(1):115-29. doi: 10.1016/j.jemermed.2014.09.007. Epub 2014 Oct 18. PMID 25440865
- [Background] Govindappagari S, Grossman TB, Dayal AK, Grosberg BM, Vollbracht S, Robbins MS. Peripheral nerve blocks in the treatment of migraine in pregnancy. Obstet Gynecol. 2014 Dec;124(6):1169-1174. doi: 10.1097/AOG.0000000000000555. PMID 25415168
- [Background] Lipton RB, Baggish JS, Stewart WF, Codispoti JR, Fu M. Efficacy and safety of acetaminophen in the treatment of migraine: results of a randomized, double-blind, placebo-controlled, population-based study. Arch Intern Med. 2000 Dec 11-25;160(22):3486-92. doi: 10.1001/archinte.160.22.3486. PMID 11112243
- [Background] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Background] James AH, Brancazio LR, Price T. Aspirin and reproductive outcomes. Obstet Gynecol Surv. 2008 Jan;63(1):49-57. doi: 10.1097/OGX.0b013e31815e8731. PMID 18081940
- [Background] Korucu O, Dagar S, Corbacioglu SK, Emektar E, Cevik Y. The effectiveness of greater occipital nerve blockade in treating acute migraine-related headaches in emergency departments. Acta Neurol Scand. 2018 Sep;138(3):212-218. doi: 10.1111/ane.12952. Epub 2018 May 10. PMID 29744871
- [Background] Allen SM, Mookadam F, Cha SS, Freeman JA, Starling AJ, Mookadam M. Greater Occipital Nerve Block for Acute Treatment of Migraine Headache: A Large Retrospective Cohort Study. J Am Board Fam Med. 2018 Mar-Apr;31(2):211-218. doi: 10.3122/jabfm.2018.02.170188. PMID 29535237
- [Background] Negro A, Delaruelle Z, Ivanova TA, Khan S, Ornello R, Raffaelli B, Terrin A, Reuter U, Mitsikostas DD; European Headache Federation School of Advanced Studies (EHF-SAS). Headache and pregnancy: a systematic review. J Headache Pain. 2017 Oct 19;18(1):106. doi: 10.1186/s10194-017-0816-0. PMID 29052046
- [Background] Schoen JC, Campbell RL, Sadosty AT. Headache in pregnancy: an approach to emergency department evaluation and management. West J Emerg Med. 2015 Mar;16(2):291-301. doi: 10.5811/westjem.2015.1.23688. Epub 2015 Feb 25. PMID 25834672
- [Background] Lipton RB, Diener HC, Robbins MS, Garas SY, Patel K. Caffeine in the management of patients with headache. J Headache Pain. 2017 Oct 24;18(1):107. doi: 10.1186/s10194-017-0806-2. PMID 29067618
- [Background] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019 May;39(6):687-710. doi: 10.1177/0333102419828967. Epub 2019 Feb 26. PMID 30806518
- [Derived] Bushman ET, Blanchard CT, Cozzi GD, Davis AM, Harper L, Robbins LS, Jones B, Szychowski JM, Digre KB, Casey BM, Tita AT, Sinkey RG. Occipital Nerve Block Compared With Acetaminophen and Caffeine for Headache Treatment in Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2023 Nov 1;142(5):1179-1188. doi: 10.1097/AOG.0000000000005386. Epub 2023 Sep 28. PMID 37769308

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (4.8) | 27.3 (5.3) | 27.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black, Non-Hispanic | 15 | 22 | 37
  Race: Hispanic | 2 | 3 | 5
  Race: White, Non-Hispanic | 14 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
BMI at Randomization [Mean (Standard Deviation); unit: kg/m^2] | 36.4 (10.5) | 37.2 (10.7) | 36.8 (10.5)
Insurance Status [Count of Participants; unit: Participants]
  None/Self-pay | 2 | 1 | 3
  Public | 17 | 26 | 43
  Private | 12 | 4 | 16
Nulliparous [Count of Participants; unit: Participants] — If the patient has never had a live birth before.
  Participants | 6 | 8 | 14
Tobacco Use [Count of Participants; unit: Participants] | 4 | 4 | 8
Marijuana Use [Count of Participants; unit: Participants] | 2 | 2 | 4
Other Illicit Substance Use [Count of Participants; unit: Participants] | 1 | 0 | 1
Gestational Age at randomization (weeks) [Mean (Standard Deviation); unit: weeks] | 28.2 (8.3) | 27.2 (7.5) | 27.7 (7.9)
Chronic Hypertension [Count of Participants; unit: Participants] | 9 | 4 | 13
Diabetes [Count of Participants; unit: Participants] | 6 | 3 | 9
Headache prior to pregnancy [Count of Participants; unit: Participants] | 12 | 18 | 30
Known primary headache disorder [Count of Participants; unit: Participants]
  Overall | 9 | 14 | 23
  Migraine | 8 | 12 | 20
  Tension | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Occipital Nerve Block in Pregnancy
Description: Based on guidelines from the International Headache Society the primary outcome is the portion of women who experience resolution of headache or improvement of headache to mild range (VRS ≤ 3) at 2 hours following treatment with Occipital nerve block as compared to acetaminophen/caffeine cocktail.
Time Frame: 60-300 min
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 20 | 16
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.30, Chi-squared

2. Secondary Outcome: Response to Treatment Within 2 Hours
Description: Visual/verbal Rating Score (VRS). VRS is used to assess pain in patients. With 0 representing no pain at all and 10 representing worst possible pain.
  Total Minimum score=0 Total Maximum score=10
  Higher values represent worse pain. If VRS=0, then the headache pain is considered resolved.
Time Frame: 2 hrs
Population: If headache was significantly improved at 1 hour, patient could leave prior to VRS at 2 hours (n=28 total patients). One patient was delivered following ONB instead of discharged due to decision for delivery prior to VRS at 2 hrs.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 13 | 20
score on a scale | 6.0 [4.0 to 8.0] | 6.5 [2.5 to 8.0]
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney) — The p-value was calculated using a 2 sided Wilcoxon rank sum test

3. Secondary Outcome: Number of Participants With Need for Crossover Treatment
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 9 | 14
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.19, Chi-squared

4. Secondary Outcome: Response to Cross Over Treatment at 60 Min
Description: as for outcome 2
Time Frame: 60 min
Population: Patients who received crossover treatment. 2 patients in the ONB did not receive crossover as they were with drawn from the study due to decision for delivery. 1 patient in the SC group declined crossover.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 9 | 14
score on a scale | 6 [4 to 8] | 3 [0 to 4]
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Need for Second Line Treatment
Time Frame: 120 min
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 5 | 5
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 1.00, Fisher Exact — P-value was calculated

6. Secondary Outcome: Response to Second Line Treatment at 60 Min
Description: as for outcome 2
Time Frame: 180min
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 5 | 5
score on a scale | 6 [4 to 7] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Participants With Need for Neurology Consult
Time Frame: 5 hours
Population: Patients with a refractory headache. Refractory headache = VRS score of >3 2 hours after second-line treatment. This prompted Neurology consultation.
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 4 | 3
Participants | 4 | 2
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.43, Fisher Exact

8. Secondary Outcome: Number of Participants With Need for Admission for Treatment of Headache
Time Frame: 7 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Need for Representation for Treatment of Headache With 28 Days
Description: Emergency department for treatment of headache since treatment asked at 28 day follow up
Time Frame: 28 days
Population: Patients who responded to specific question at 28 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 24 | 23
Participants | 5 | 1
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.19, Fisher Exact

10. Secondary Outcome: Number of Participants With Development of Hypertensive Disease of Pregnancy Within 28 Days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 9 | 4
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.18, Fisher Exact

11. Secondary Outcome: Number of Participants With Satisfaction of Response Treatment at 7 Days
Time Frame: 7 days
Population: Patients who responded to specific question at 7 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 23 | 23
Participants
  Strongly satisfied | 12 | 10
  Satisfied | 5 | 4
  Neutral | 3 | 5
  Dissatisfied | 1 | 1
  Very dissatisfied | 2 | 3
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.92, Fisher Exact

12. Secondary Outcome: Duration of Headache Free Period at 7 Days
Time Frame: 7 days
Population: Patients who responded to specific question at 7 day follow up.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 14 | 18
days | 6 [0.5 to 7] | 1 [0 to 5]
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number of Participants With Development of Hypertensive Disease of Pregnancy Within 7 Days
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 31 | 31
Participants | 7 | 2
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.14, Fisher Exact

14. Secondary Outcome: Number of Participants With Injection Site Complication (Infection, Hematoma, and Ecchymosis)
Description: Other: Pain at injection site
Time Frame: 7 days
Population: Number of patients who responded to specific question at 7 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
Number analyzed (Participants) | 24 | 23
Participants | 0 | 2
Statistical Analysis 1: Comparison: Occipital Nerve Block vs Oral Acetaminophen/Caffeine Group; Test type: Superiority; p = 0.23, Fisher Exact

ADVERSE EVENTS:
Time Frame: Occurring within 28 days of treatment.
Arm/Group | Occipital Nerve Block | Oral Acetaminophen/Caffeine Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Occipital Nerve Block (N=31) | Oral Acetaminophen/Caffeine Group (N=31)
Pre-term Birth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — PTB, Sev SiPreE, not related to study
Injection Site Complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Patients reported pain at injection site of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03951649/Prot_SAP_000.pdf